CLINICAL TRIAL: NCT03987256
Title: Tennis Elbow, Randomized Study: Needling With and Without Platelet-rich Plasma After Failure of Up-to-date Rehabilitation
Brief Title: ECRB Tendinopathy: Needling ± PRP After Failure of Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Adrien Schwitzguebel (Other)
Responsible Party: Sponsor-Investigator, Adrien Schwitzguebel, Independent physician, Hôpital de la Providence, Switzerland
Organization: Hôpital de la Providence, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECRB_Conservative
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Tennis Elbow; PRP; Tendinopathy; Tendinosis; Extracorporal Shockwave Therapy (ESWT); Tendon Needling (Peppering); Extensor Carpi Radialis Brevis (ECRB)
Keywords: tennis elbow; PRP; Focussed shockwave therapy; needling; tendinopathy
MeSH Terms: conditions — Tennis Elbow; Tendinopathy | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: In both groups, needling will be performed. Half of the patients will receive PRP (platelet-rich plasma).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients will have blood puncture. Then, the research coordinator will prepare either an opaque syringe of saline solution or of PRP. At the end of the needling procedure, the investigator will inject the content of the opaque syringe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECRB needling with adjuvant PRP infiltration (Experimental): First step: rehabilitation protocol during 3 months including focal shockwave therapy
  Second step: one single tendon needling with PRP
  Interventions: Other: Initial rehabilitation protocol; Procedure: Needling with PRP
- ECRB needling with adjuvant NaCl 0.9% infiltration (Active Comparator): First step: rehabilitation protocol during 3 months including focal shockwave therapy
  Second step: one single tendon needling with Saline solution
  Interventions: Other: Initial rehabilitation protocol; Procedure: Needling with saline solution

INTERVENTIONS:
Other: Initial rehabilitation protocol — During 12 weeks, under kinesitherapist guidance, patients will perform daily eccentric stretching and strengthening of the ECRB and periscapular musculature, manual therapies, and kinesiotaping. They will also use orthotics after 6 weeks if kinesiotaping is not effective. At weeks 1-5, patients will undergo weekly ultrasound-guided focused shockwave therapy under the following protocol: 0,15- 0,30mJ/mm2 (the highest energy flux the patient can well tolerate), 1500 shocks at 5Hz at the origin of common extensor or flexor tendon.
Procedure: Needling with PRP — In case of failure of proper rehabilitation and shockwave therapy, patients will have a block of the radialis nerve just above the arcade of Frohse with 1 ml of procaine 2%. Then, a single needling of the ECRB enthesis (peppering technique) will be performed as follow: , ultrasound-guided, 25 repetitions with a 20 gauge needle. At the end of the procedure, the lesion will be fulfilled with PRP.
  Details of PRP preparation (ACP Arthrex): 15 ml of blood, no activators or anticoagulants, poor in white blood cells (the last mm of buffy coat above the red blood cells pellet is not collected).
  Excentric stretching and strengthening, as well as orthotics or kinesiotaping will be continued as long as symptoms persists during the 6 first months after the needling procedure.
  Arms: ECRB needling with adjuvant PRP infiltration
Procedure: Needling with saline solution — In case of failure of proper rehabilitation and shockwave therapy, patients will have a block of the radialis nerve just above the arcade of Frohse with 1 ml of procaine 2%. Then, a single needling of the ECRB enthesis (peppering technique) will be performed as follow: , ultrasound-guided, 25 repetitions with a 20 gauge needle. At the end of the procedure, the lesion will be fulfilled with saline solution.
  Excentric stretching and strengthening, as well as orthotics or kinesiotaping will be continued as long as symptoms persists during the 6 first months after the needling procedure.
  Arms: ECRB needling with adjuvant NaCl 0.9% infiltration

SUMMARY:
This study evaluates the effect of platelet-rich plasma (PRP) use during needling of the extensor carpalis radialis brevis tendon, after failure of proper reeducation including focal extra-corporal shockwave therapy (ESWT). Half of the patients with receive PRP and needling, and half of the patients will receive needling alone.

During the reeducation, the clinical evaluation will be monitored and reported as in a case series.

DETAILED DESCRIPTION:
The conservative management of lateral epicondylitis is known to be a difficult-to-treat annoying condition. The first-line conservative management includes physical therapies with adjuvant painkillers and orthotics, and usually extracorporal shockwave therapy (ESWT). In clinical practice, infiltrative therapies a performed either before or after shockwave therapies. In the author's point of view, they represent a second-line conservative treatment.

The success rate of ESWT for lateral epicondylitis depends mainly of the protocol used. Especially, poor results were observed with too low energy. Both radial and focal ESWT are effective, and focal ESWT has been showed as being as effective as surgical tenotomy.

Concerning infiltrative therapies, it has been well established that corticosteroids are efficient in short-term but deleterious in long-term, likely for degenerative purposes. Prolotherapy, autologous blood, and botulinic toxin injections and others infiltrative therapies are less studied and therefore nowadays not clearly supported by the literature. Stem cells might be an alternative in the future.

Platelet-rich-plasma (PRP) is nowadays widely used, but the results of clinical trials are discordant. Even if the superiority of PRP over corticosteroids is well established, the superiority of PRP on tendon needling or peppering is still controversial. Martin et al. 2019 found in a partially blinded randomized controlled trial (RCT) involving 71 patients no clinical differences at 6 months of follow-up between 2 sessions of peppering with saline + local anesthetic and PRP + local anesthetic. In a similar unblended RCT involving 50 patients, Schöffl et al. 2017 found no clinical differences at 6 months of follow-up. Montalvan et al. 2016 found in a RCT involving 50 patients between 2 infiltrations of PRP and saline no clinical differences at 6 months of follow-up. Rehabilitation was not allowed during the trial and the tendon was not peppered. Mishra et al. found in a blinded RCT involving 119 patients a positive clinical effect of PRP on saline solution, using a single injection with peppering. Behera et al. found similar results in a small RCT on 25 patients.

Some factors has been advocated to influence the outcomes. The most relevant are: direct mechanic action of the needle and fenestration (peppering) technique, number of PRP injections, cells count (platelets, white blood- and red blood cells), activation of the platelets, concomitant local anesthetic use, peri-interventional use of NSAIDs and corticosteroids, concomitant rehabilitation or a contraria immobilization. Whether the positive results observed into the previous selected studies are due to either PRP, peppering, or any of the confounding factors described above remains to debate.

The first aim of this study is to determine the proportion of patients, which would need an infiltrative technique after a proper rehabilitation protocol involving physical therapies, orthotics and ESWT. Our second aim is to establish whether PRP as adjuvant therapy to peppering would increase clinical outcomes.

Details of sample size calculation (58 overall, 29 per group):

58 patients are required to have a 95% chance of detecting, as significant at the 5% level, an increase in the primary outcome measure from 50 in the control group to 60 in the experimental group, considering a standard deviation of 10% and a dropout rate of 10%. After the inclusion of 40 patients, the standard deviation will be re-evaluated and the sample size corrected accordingly if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Lesion of the ECRB tendon on ultrasonography ([hypoechogenic area during rest OR hypoechogenic area during active contraction, OR compressibility of the tendon OR doppler signal] AND [positive sonopalpation])
* Failure to rehabilitation program including shockwave therapy defined as the need for the patient undergoing additional therapies

Exclusion Criteria:

* Presence on ultrasound of an isolated lesion of the superficial epicondylar tendons as described above, with intact ECRB
* Presence on ultrasound of any of: radiohumeral synovial material; interruption of the lateral collateral ligament; radial nerve entrapment, i.e. under the arcade of Frohse; osteochondral lesion; joint effusion. Note: calcic enthesophytes are not considered as an exclusion criteria
* Clinical presence of cervicobrachialgia, or pain irradiating into the hand
* Corticosteroids: oral intake or infiltration on the last 3 months
* Proximal radius fracture history
* Active inflammatory rheumatic disorders
* Diabetes mellitus
* Immunocompromized status
* Allergy to local anesthetics
* Bleeding disorders or current anticoagulation therapy
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiopulmonary significant insufficiency, etc.)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Pain during isometric contraction of the ECRB | 3 months
  Pain is evaluated on a 0-10 scale (0 = no pain) during isometric contraction maneuver of the ECRB

SECONDARY OUTCOMES:
Pain during isometric contraction of the ECRB | -3, 0, 6, & 12 months
  Pain is evaluated on a 0-10 scale (0 = no pain) during isometric contraction maneuver of the ECRB
Overall pain evaluation (mean of the 3 last days) | -3, 0, 3, 6, & 12 months
  Pain is evaluated on a 0-10 scale (0 = no pain)
SANE score (Single Assessment Numeric Evaluation) | -3, 0, 3, 6, & 12 months
  Function is evaluated on a 0-100% scale (100 = good function)
PRTEE score (Patient-Rated Tennis Elbow Evaluation) | -3, 0, 3, 6, & 12 months
  Score going from 0 to 100 (0 = good outcome)
Strength on Jamar test (hand grip strength) | -3, 0, 3, 6, & 12 months
  Grip strength measured in Kg (Higher strength = better outcome)
Proportion of patient cured with reeducation protocol | 0 months
  Descriptive statistics: Evaluation of the proportion of patients for which the tendon needling is not necessary
Volume of PRP prepared | 0 months
  Descriptive statistics: Quantity of PRP prepared (in ml)
Volume of PRP (or saline solution) injected | 0 months
  Descriptive statistics: Quantity of PRP (or saline solution) injected (in ml)
Ultrasonographic aspect of the epicondylar tendon: Hypoechogenic lesion | -3, 0, 3, & 6 months
  The tridimensional volume of the lesion is measured in mm^3
Ultrasonographic aspect of the epicondylar tendon: Doppler | -3, 0, 3, & 6 months
  The Doppler reaction will be evaluated on a subjective scale (none, mild, average, high, huge)
Ultrasonographic aspect of the epicondylar tendon: Solution of continuity | -3, 0, 3, & 6 months
  During active contraction of the ECRB, an eventual solution of continuity will be measured in mm
Ultrasonographic aspect of the epicondylar tendon: Thickness | -3, 0, 3, & 6 months
  The thickness of the common epitrochlear will be measured in mm
Ultrasonographic aspect of the epicondylar tendon: Compressibility | -3, 0, 3, & 6 months
  The presence or absence of compressibility of the common epitrochlear tendon (binary outcome)
Ultrasonography of the epicondylar tendon: Sonopalpation | -3, 0, 3, & 6 months
  The patient pain on sonopalpation will be evaluated on a 0-10 scale (0= no pain)

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Schwitzguébel, MD, Principal Investigator — Hôpital de La Providence
Locations (1):
- Hôpital La Providence, Sports Medicine, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerdesmeyer L, Mittermayr R, Fuerst M, Al Muderis M, Thiele R, Saxena A, Gollwitzer H. Current evidence of extracorporeal shock wave therapy in chronic Achilles tendinopathy. Int J Surg. 2015 Dec;24(Pt B):154-9. doi: 10.1016/j.ijsu.2015.07.718. Epub 2015 Aug 29. PMID 26327530
- [Background] Park JW, Hwang JH, Choi YS, Kim SJ. Comparison of Therapeutic Effect of Extracorporeal Shock Wave in Calcific Versus Noncalcific Lateral Epicondylopathy. Ann Rehabil Med. 2016 Apr;40(2):294-300. doi: 10.5535/arm.2016.40.2.294. Epub 2016 Apr 25. PMID 27152280
- [Background] Coombes BK, Bisset L, Vicenzino B. Efficacy and safety of corticosteroid injections and other injections for management of tendinopathy: a systematic review of randomised controlled trials. Lancet. 2010 Nov 20;376(9754):1751-67. doi: 10.1016/S0140-6736(10)61160-9. Epub 2010 Oct 21. PMID 20970844
- [Background] Houck DA, Kraeutler MJ, Thornton LB, McCarty EC, Bravman JT. Treatment of Lateral Epicondylitis With Autologous Blood, Platelet-Rich Plasma, or Corticosteroid Injections: A Systematic Review of Overlapping Meta-analyses. Orthop J Sports Med. 2019 Mar 14;7(3):2325967119831052. doi: 10.1177/2325967119831052. eCollection 2019 Mar. PMID 30899764
- [Background] Gautam VK, Verma S, Batra S, Bhatnagar N, Arora S. Platelet-rich plasma versus corticosteroid injection for recalcitrant lateral epicondylitis: clinical and ultrasonographic evaluation. J Orthop Surg (Hong Kong). 2015 Apr;23(1):1-5. doi: 10.1177/230949901502300101. PMID 25920633
- [Background] Dong W, Goost H, Lin XB, Burger C, Paul C, Wang ZL, Kong FL, Welle K, Jiang ZC, Kabir K. Injection therapies for lateral epicondylalgia: a systematic review and Bayesian network meta-analysis. Br J Sports Med. 2016 Aug;50(15):900-8. doi: 10.1136/bjsports-2014-094387. Epub 2015 Sep 21. PMID 26392595
- [Background] Sims SE, Miller K, Elfar JC, Hammert WC. Non-surgical treatment of lateral epicondylitis: a systematic review of randomized controlled trials. Hand (N Y). 2014 Dec;9(4):419-46. doi: 10.1007/s11552-014-9642-x. PMID 25414603
- [Background] Lai WC, Erickson BJ, Mlynarek RA, Wang D. Chronic lateral epicondylitis: challenges and solutions. Open Access J Sports Med. 2018 Oct 30;9:243-251. doi: 10.2147/OAJSM.S160974. eCollection 2018. PMID 30464656
- [Background] Imam MA, Holton J, Horriat S, Negida AS, Grubhofer F, Gupta R, Narvani A, Snow M. A systematic review of the concept and clinical applications of bone marrow aspirate concentrate in tendon pathology. SICOT J. 2017;3:58. doi: 10.1051/sicotj/2017039. Epub 2017 Oct 9. PMID 28990575
- [Background] Mi B, Liu G, Zhou W, Lv H, Liu Y, Wu Q, Liu J. Platelet rich plasma versus steroid on lateral epicondylitis: meta-analysis of randomized clinical trials. Phys Sportsmed. 2017 May;45(2):97-104. doi: 10.1080/00913847.2017.1297670. Epub 2017 Mar 3. PMID 28276986
- [Background] Martin JI, Atilano L, Merino J, Gonzalez I, Iglesias G, Areizaga L, Bully P, Grandes G, Andia I. Platelet-rich plasma versus lidocaine as tenotomy adjuvants in people with elbow epicondylopathy: a randomized controlled trial. J Orthop Surg Res. 2019 Apr 23;14(1):109. doi: 10.1186/s13018-019-1153-6. PMID 31014382
- [Background] Schoffl V, Willauschus W, Sauer F, Kupper T, Schoffl I, Lutter C, Gelse K, Dickschas J. Autologous Conditioned Plasma Versus Placebo Injection Therapy in Lateral Epicondylitis of the Elbow: A Double Blind, Randomized Study. Sportverletz Sportschaden. 2017 Jan;31(1):31-36. doi: 10.1055/s-0043-101042. Epub 2017 Feb 21. PMID 28222465
- [Background] Montalvan B, Le Goux P, Klouche S, Borgel D, Hardy P, Breban M. Inefficacy of ultrasound-guided local injections of autologous conditioned plasma for recent epicondylitis: results of a double-blind placebo-controlled randomized clinical trial with one-year follow-up. Rheumatology (Oxford). 2016 Feb;55(2):279-85. doi: 10.1093/rheumatology/kev326. Epub 2015 Sep 8. PMID 26350485
- [Background] Mishra AK, Skrepnik NV, Edwards SG, Jones GL, Sampson S, Vermillion DA, Ramsey ML, Karli DC, Rettig AC. Efficacy of platelet-rich plasma for chronic tennis elbow: a double-blind, prospective, multicenter, randomized controlled trial of 230 patients. Am J Sports Med. 2014 Feb;42(2):463-71. doi: 10.1177/0363546513494359. Epub 2013 Jul 3. PMID 23825183
- [Background] Behera P, Dhillon M, Aggarwal S, Marwaha N, Prakash M. Leukocyte-poor platelet-rich plasma versus bupivacaine for recalcitrant lateral epicondylar tendinopathy. J Orthop Surg (Hong Kong). 2015 Apr;23(1):6-10. doi: 10.1177/230949901502300102. PMID 25920634
- [Background] Kaux JF, Emonds-Alt T. The use of platelet-rich plasma to treat chronic tendinopathies: A technical analysis. Platelets. 2018 May;29(3):213-227. doi: 10.1080/09537104.2017.1336211. Epub 2017 Jul 31. PMID 28759287
- [Derived] Schwitzguebel AJ, Bogoev M, Nikolov V, Ichane F, Ladermann A. Tennis elbow, study protocol for a randomized clinical trial: needling with and without platelet-rich plasma after failure of up-to-date rehabilitation. J Orthop Surg Res. 2020 Oct 7;15(1):462. doi: 10.1186/s13018-020-01998-8. PMID 33028383